CLINICAL TRIAL: NCT02877446
Title: Observatoire Des Assistances Monoventriculaires Gauches du Grand Sud
Brief Title: South Of France Cardiac Assist Registry
Acronym: SOFCAR
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: University Hospital, Toulouse (Other); University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: 9690
Record Dates: First submitted 2016-07-08; First posted 2016-08-24 (Estimated); Last update posted 2022-08-11 (Actual); Status verified 2022-04

CONDITIONS: Chronic or Acute Advanced Heart Failure
Keywords: Left ventricular assist device (LVAD); Terminal heart failure; Ventricular assist device (VAD)
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Chronic heart failure is a common disease. It is also a serious disease with a mortality of 50% at 5 years, representing a significant cost in terms of public health expenditure.

Heart transplantation represents the "gold standard" of care for terminal heart failure patients reached the end of the disease despite optimal medical and surgical management of their disease, with a survival rate of transplant patients by 90% at 1 year and 82% at 3 years.

Long term LVAD are an innovative technology available for more than a decade, developed in part because of the shortage of cardiac grafts and high mortality among patients waiting for transplants due to an important pending.

This technique is used substantially only for ten to fifteen years in the world. Survival after implantation of latest devices reaches 80% at 1 year.

In France, this technique is intended for patients with terminal heart failure who ended different pharmacological and invasive therapeutic resources available.

Currently, academic centers that offer the possibility of long-term LVAD support are organized unicentric in order to centralize specialized care for these patients.

Indeed, patients candidates for the establishment of a long-term LVAD are rigorously selected to ensure an acceptable survival.

However, practices vary considerably from one center to another in particular regarding:

* Implantation indications,
* Pre-implantation patient assessment,
* Monitoring,
* Implementation of pharmacological treatments, particularly anticoagulants or betablockers.

DETAILED DESCRIPTION:
Methods:

It's a prospective multicentric observational study realised on 3 University Hospital in France: Bordeaux, Montpellier and Toulouse.

Population:

All patients undergoing implantation of a long-term LVAD support whatever the brand and type, on one of the 3 participating centers (Montpellier, Toulouse or Bordeaux) during the 3 years period, after approval of informed consent.

Patients were followed up at 1 and 6 months, and 1 year as part of their routine management of their disease.

Patients should have agreed to participate in the observatory, knowing that participation or refusal to participate will not alter the therapeutic attitude of the team responsible for the patient.

Aim:

Main aim is 1 year mortality of LVAD recipients

Secondary aim are:

* Descriptive epidemiology of LVAD implantation: prevalence, etiology, affected populations
* Description of the state of practice: indications, against-indications, preimplantation data, intraoperative data, postoperative data, tracking data
* Rating prognosis of patients under LVAD support
* In-hospital, 30 days, 6 months, and 1 year survival
* Number of transplanted and assisted patients at 1 year
* Evaluation of complications (infections, bleeding, thromboembolism, equipment failures, ...)
* Analyses in subgroups according to age, sex, initial indication (including ischemic heart disease vs nonischemic), assistance used and year of implantation
* Research of prognostic factors for postoperative and chronic right ventricular failure, prognostic factors of cardiovascular and all causes death.

Feasibility:

Based on historical data of the concerned centers (CHU Montpellier, Bordeaux and Toulouse) and recent predictions of french health authority HAS ("Haute Autorité de Santé"), 200 patients are provided in the observatory register, rhythm about 20-30 patients per year per center for a 3-year recruitment period Monitoring will be carried out by the referring physician for each patient at 1 and 6 months, and at 1 year in the usual care of pathology in each center with the possibility to adapt the follow-up date to +/- 1 month.

For patients who have moved and have therefore changed of referral center, an evaluation at one year will be made by mail or phone contact with the physician and / or patient.

Collect and circulation of patients' data:

Data will be collected under the patient's referring physician's responsibility in each center. Data will be entered directly into the electronic database (e-CRF) developed University of Montpellier.

Patient will be identified by the number of the center (1 = Bordeaux, 2 = Montpellier 3 = Toulouse) followed by the first letter of the name and the first initial and the center of the patient number in question (automatic chronological number according to the entry on the e-CRF - data coding is integrated into the e-CRF) Monitoring at 1 month, 6 months and 1 year, will be completed by the middle of referring physicians and entered directly into the electronic database.

There will be no traffic data on paper for these two steps.

In case of lost sight, follow-up at 1 year will be carried out by the centers, by phone or mail from the municipality of birth, the attending physician or cardiologist and patient, which requires knowledge of the date full birth patients to avoid confusion.

For the analysis, data will be anonymized (as shown above).

Members of the scientific committee, persons responsible for logistics and coordination statistics will have access to all of the identified data.

Research data is entered via an electronic case report forms (e-CRF) developed from the Capture System software (CLINSIGHT company), enabling quality control of data in real time. To meet regulatory requirements, this software complies with the FDA's recommendations on Computerized Systems for Managing Clinical Trials and electronic signature and standards (CDISC, ICH, GCP 2001/20 / EC ...). The connection is via a password and a unique identifier specific to each user that will give access only to his patients himself. An audit function is integrated allowing traceability of data as well as changes. The encrypted data will then be transmitted to the responsible center of the data-management via a secure internet connection.

The e-CRF must be composed of all the information required by the protocol.

Information and Consent of participants:

Prior to the completion of this research, the free, writing and informed consent of patients must be collected after information by the investigator during a consultation, and after a sufficient period of reflection.

Participants information for research should be written simply, in language understandable by the patient. After having read the participant and the investigator will have dated and signed the consent form (original archived by the investigator and an original will be given to research participants).

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing implantation of LVAD support whatever make and type on one of the 3 participating centers (University Hospital of Montpellier, Toulouse and Bordeaux) during the period
* Free, informed and signed consent
* Adults
* Men or women Patients should have agreed to participate in the observatory, knowing that participation or refusal to participate will not alter the therapeutic attitude of the physician responsible for the patient. Study of phenotypic characteristics will not change the therapeutic approach of the medical teams.

Exclusion Criteria:

* Patient unable to understand the nature and goals of the study and / or communication difficulties with the investigator
* Major protected by law (guardianship, curatorship or under judicial protection)
* Patient deprived of liberty by judicial or administrative decision

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent surgical LVAD implantation in one of the 3 participating centers (University Hospital of Montpellier, Toulouse and Bordeaux, France) for a period of 3 years, will be consecutively included whatever type of LVAD (Heartmate 2 or 3®, Jarvik®, Heartware®,…).
  Patients will be follow-up at 1 and 6 months, and 1 year. Patients should have agreed to participate in the observatory, knowing that participation or refusal to participate will not alter the therapeutic attitude of the physician responsible for the patient. Study of phenotypic characteristics will not change therapeutic approach of the medical teams.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2022-04 (Actual); Study Completion 2022-08-10 (Actual)

PRIMARY OUTCOMES:
Mortality rate | 1 year
  Mortality rate after one year for patients included in the research

SECONDARY OUTCOMES:
Cardiovascular death rates | 30 days
  Search prognostic factors for postoperative ventricular failure and chronic right, prognostic factors of cardiovascular death and all-cause
Cardiovascular death rates | 6 months
  Search prognostic factors for postoperative ventricular failure and chronic right, prognostic factors of cardiovascular death and all-cause
Cardiovascular death rates | 1 year
  Search prognostic factors for postoperative ventricular failure and chronic right, prognostic factors of cardiovascular death and all-cause
Mortality rate | 30 days
Mortality rate | 6 months
vital function | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Francois Roubille, MD PHD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- University Hospital of Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
ND